CLINICAL TRIAL: NCT00510744
Title: Pancreatic Enzymes to Restore Digestive Function in Malnourished Gastric Bypass Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Stephen O'Keefe, Professor of Medicine, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO07070305
Record Dates: First submitted 2007-08-01; First posted 2007-08-02 (Estimated); Results first posted 2016-06-02 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-04

CONDITIONS: Obesity
Keywords: obesity, bariatric surgery, pancreatic secretion
MeSH Terms: conditions — Obesity | interventions — Pancrelipase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pancreatic enzyme supplementation (Experimental): 3 month supplementation in those gastric bypass patients shown to have a fat absorption less than 80%
  Interventions: Drug: pancreatic enzyme supplement

INTERVENTIONS:
Drug: pancreatic enzyme supplement — 4 caps with meals, 2 with snacks
  Other Names: Creon

SUMMARY:
Hypothesis: Bypass of the upper GI tract with bariatric surgery results in suppression of pancreatic function resulting in maldigestion and further malabsorption. In this study we will measure pancreatic secretion in previously obese gastric bypass patients with excessive weight loss. If malabsorption is associated with diminished pancreatic secretion, we will test over a 3 month period whether supplementation with enzyme supplements prevent further weight loss.

DETAILED DESCRIPTION:
Obesity has reached epidemic proportions in the USA and Europe, and is increasing world-wide. Morbid obesity (BMI>40kg/m2) is usually resistant to medical and dietary therapy while surgical treatment results in a permanent loss of most of the excess weight. The most popular technique today is the Roux-en-Y gastric bypass procedure which results in a weight loss of approximately 95 lbs per year or a 2/3 loss of the excess weight in 2 years (7-9). Weight loss occurs for 2 reasons: first the volume of the stomach is reduced, and second, the duodenum and first part of the jejunum is bypassed resulting in malabsorption. Although most patients tolerate the procedure well with a leveling off of weight loss close to the ideal body weight, a subpopulation of patients continue to lose weight, becoming progressively more malnourished, necessitating reversal of the surgery. To date, no studies have investigated what happens to pancreatic function in obese patients following bypass surgery, but from an understanding of the physiology of pancreatic stimulation, it is likely that the pancreas atrophies because the intestinal phase of pancreatic stimulation is bypassed and the inhibitory ileal brake is perpetually stimulated. In the following study we plan to investigate whether patients with excessive weight loss after bypass surgery develop malabsorption not only due to bypass of the upper GI tract but also because of impaired pancreatic enzyme secretion resulting from chronic activation of the ileal brake mechanism. Up to 20 post-bariatric surgery (Roux-en-Y) patients with excessive and continued weight loss will be screened for fat absorption and loss of pancreatic secretion. Those with loss of >20% fat absorption will then be treated at home with pancreatic enzyme supplements for a 3 month period to assess weight stabilization or gain. After 3 months, fat absorption and the pancreatic stimulation test will be repeated while patients are on enzyme supplementation to determine whether fat digestion and absorption has improved from baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults >18yrs
2. h/o Roux-en-Y gastric bypass procedure
3. Pre-surgery BMI >40Kg/m2
4. Weight loss of >30%, or 100lbs in 1st year following bypass surgery
5. Able to consume normal requirement levels of food. This will be determined from history (see above) and confirmed during the 72h food-balance study in the GCRC.

Exclusion Criteria:

1. Chronic pancreatic disease as evidenced by history, pancreatic imaging (CT or MRP scanning or ERCP) or alcohol abuse (>3 units of alcohol/day) as documented by family or care givers
2. h/o intestinal resection other than gastric bypass
3. Unstable cardio-respiratory status (BP diastolic >100mmHg, systolic >200 or <80 mmHg), ambient pO2 <90%
4. Presence of chronic inflammatory bowel or chronic small intestinal mucosal disease confirmed by radiology and biopsy.
5. Current history of feeding disorder, such as bulimia nervosa. This will be excluded by the interview and attestation of spouses, close relatives, or home companions
6. Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-08; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J O'Keefe, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh GCRC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
with publication

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pancreatic Enzyme Supplementation
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pancreatic Enzyme Supplementation
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 49 [22 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Fat Absorption
Description: 72 hour fat absorption study
Time Frame: 3 months
Population: each patients as their own control, baseline fat absorption vs post 3 month enzyme supplementation fat absorption
Measure: Mean (Standard Error); unit: g/d
Groups:
- Pancreatic Enzyme Supplementation: 3 month supplementation in those gastric bypass patients shown to have a fat absorption less than 80%
  The ability of pancreatic enzyme supplement: 4 caps with meals, 2 with snacks to improve fat absorption
Arm/Group | Pancreatic Enzyme Supplementation
Number analyzed (Participants) | 5
g/d | 60.6 (13.4)
Statistical Analysis 1: Comparison: Pancreatic Enzyme Supplementation; paired changes in fat absorption assessed by parametric (t test) or non-parametric tests (Mann-Whitney); Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.2, Standard Error of Mean 24

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Pancreatic Enzyme Supplementation
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes